CLINICAL TRIAL: NCT04642521
Title: Anaemia and Handgrip Strength, a Prospective Observatonal Study Amongst Female Population Planned for Major Elective Surgery
Brief Title: Association Between Anaemia and Handgrip Strength in Female Planned for Major Surgery and the Effect of Intravenous Iron on Handgrip Strength
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Other Study IDs: Anaemiahandgrip
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Anemia; Iron-deficiency; Patient Blood Management; Iron Deficiency Anemia
Keywords: handgrip strength; intravenous iron
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iron deficiency anaemia: Preoperatively, participants who are iron deficient with or without anaemia will receive intravenous iron (Monofer) as per ProPBM protocol.
  Interventions: Device: Jamar hydraulic hand dynamometer
- No iron deficiency anaemia: Patient in this group will not be given intravenous iron.
  Interventions: Device: Jamar hydraulic hand dynamometer

INTERVENTIONS:
Device: Jamar hydraulic hand dynamometer — The strength of the dominant hand will be recorded before and after receiving intravenous iron.
  Each participant will be positioned in a straight back chair with both hand and feet flat on the ground, elbow flexed to 90 degrees with forearm and wrist in the neutral position. Patient's muscle strength will then be tested three times with an interval of one minute between testing and the average of three times will be recorded to the nearest 0.1kg.
  Other Names: Handgrip strength

SUMMARY:
This is a sub-study parallel to ProPBM : A Randomised Control Trial Comparing a Modified Patient Blood Management Protocol Against Standard Care for Patients Undergoing Major Surgery (NCT03888768).

Only female participants of ProPBM will be included in this sub-study.

Association between anaemia and handgrip strength and the effect of intravenous iron therapy as part of ProPBM protocol within female participants is elucidated in this study.

DETAILED DESCRIPTION:
BACKGROUND:

Maximal physical efforts and aerobic exercise depend highly on adequate oxygen supply provided by haemoglobin and level of iron bound to haemoglobin.

Handgrip strength has been shown to have a strong validity and high reliability in testing the upper body and lower body muscle strength, however its use as a potential tool to identify early anaemic patients planned for surgery is not fully explored. To our knowledge, this study is the first to investigate the diagnostic power of functional performance test within preoperative anaemic population and the change of handgrip strength after administration of intravenous iron.

METHODS:

At recruitment of ProPBM study, all eligible patients for this sub-study will be invited to this sub-study and have their full blood count, ferritin and transferrin saturation recorded and handgrip strength assessed.

After randomization, those within the ProPBM protocol will receive IV iron therapy as indicated. Participants who are randomized to standard care will follow usual medical management.

Participants will be admitted 1 day prior to surgery. On admission, preoperative bloods and handgrip strength will be repeated for patients who were randomized into the ProPBM arm.

ELIGIBILITY:
Inclusion Criteria:

* Female patients participating in the ProPBM study
* Undergoing major surgery in gynaecology, gastrointestinal surgery and orthopaedics surgery
* The patient must be willing and able to provide informed consent for the study

Exclusion Criteria:

* Patients with known muscle weakness eg myasthenia gravis
* Patients with cerebrovascular or orthopaedic disease that could influence muscle mass and/or upper body function
* Patients in which IV iron is contraindicated eg 1st trimester of pregnancy or known allergy or hypersensitivity to parenteral iron
* Patients with iron overload

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female population
Study Population: Female participants of ProPBM study who are planned for major elective surgery, both anaemic and non anaemic patients are included
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-11-18 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Association between handgrip strength and haemoglobin status within female participants of ProPBM study | At recruitment
  The dependent variable is concentration of plasma circulating haemoglobin (Hb) taken at recruitment and measured in g/dL.
  The non-dependant variable is the baseline handgrip strength recorded in kilogram using Jamar hydraulic hand dynamometer. Participants will be positioned in a straight back chair with both hand and feet flat on the ground, elbow flexed to 90 degrees with forearm and wrist in the neutral position. Patient's muscle strength will then be tested three times with an interval of one minute between testing and the average of three times will be recorded to the nearest 0.1kg.
  The association between anaemia and handgrip strength will be analyzed by using binary logistic regression technique.

SECONDARY OUTCOMES:
Association between handgrip strength and iron status within female participants of ProPBM study | At recruitment
  Iron status is measured by ferritin level (mcg/L) and transferrin saturation (percentage value).
  Association between iron status and handgrip strength will be analysed using a linear regression technique.
Change in handgrip strength in iron deficient female participants of ProPBM study who received intravenous iron | Handgrip strength repeated within 1 month post IV iron administration preoperatively
  Participants who received intravenous iron will have their ferritin level, TSAT and handgrip strength reassesed during preoperative admission.
  Handgrip strength after IV iron administration will be compared to baseline handgrip strength.

CONTACTS AND LOCATIONS:
Overall Officials: Ina I Shariffuddin, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistic analysis plan

REFERENCES:
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Joosten E, Detroyer E, Milisen K. Effect of anaemia on hand grip strength, walking speed, functionality and 1 year mortality in older hospitalized patients. BMC Geriatr. 2016 Aug 19;16(1):153. doi: 10.1186/s12877-016-0326-y. PMID 27543049
- [Result] Santos PHS, Carmo EA, Carneiro JAO, Nery AA, Casotti CA. Handgrip strength: An effective screening instrument for anemia in the elderly women. Public Health Nurs. 2019 Mar;36(2):178-183. doi: 10.1111/phn.12579. Epub 2019 Jan 9. PMID 30628133